CLINICAL TRIAL: NCT04531696
Title: UZ/KU Leuven Program for Post-mortem Tissue Donation to Enhance Research
Acronym: UPTIDER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other); Universiteit Antwerpen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: S64410
Record Dates: First submitted 2020-08-11; First posted 2020-08-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer; Hereditary Diseases
MeSH Terms: conditions — Breast Neoplasms; Genetic Diseases, Inborn | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard (Other): UPTIDER consists of 8 substudies:
  1. Pilot phase
  2. Invasive Lobular Carcinoma (ILC) substudy
  3. Inflammatory Breast Cancer (IBC) substudy
  4. Molecular heterogeneity and treatment response substudy
  5. Patient-derived xenograft (PDX) / Patient-derived Organoid (PDO) substudy
  6. Metabolomics substudy
  7. Liquid biopsy substudy
  8. Hereditary cancer syndromes substudy The intervention, consisting of sample collection only, is identical in all substudies, however, the focus of downstream analysis of the samples may be different.
  Interventions: Procedure: Blood draw; Procedure: Post-mortem tissue collection

INTERVENTIONS:
Procedure: Blood draw — Blood draw at inclusion
Procedure: Post-mortem tissue collection — Sample collection (both liquids, tumour tissue and non-tumour tissue) during post-mortem research autopsy

SUMMARY:
UPTIDER is a prospective, interventional, non-Investigational Medicinal Product (non-IMP), non-commercial, single centre post-mortem tissue donation program for metastatic breast cancer patients or patients with a germline pathogenic variant with a moderate to high lifetime risk of breast cancer and at least one malignancy at time of death. The overarching objective of UPTIDER is (i) to unravel metastatic breast cancer evolution, biology, heterogeneity and treatment resistance and (ii) to assess pathogenicity and tumour biology in hereditary cancer syndromes with a high lifetime risk of breast cancer; both through extensive post-mortem multi-level and multi-region sample analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Signature of informed consent by the subject.
* Metastatic breast cancer, or hereditary cancer syndrome with a moderate to high lifetime risk of breast cancer, for which the patient is treated/followed in UZ Leuven or treated in another hospital and referred to UZ Leuven specifically for the trial.

Additional inclusion criteria for the different substudies:

* Pilot phase: no additional inclusion criteria.
* ILC substudy: histologically confirmed history of ILC.
* IBC substudy: history of IBC, fulfilling the following criteria described by Dawood et al: rapid onset of breast erythema, oedema and/or peau d'orange and/or warm breast with or without an underlying palpable mass, duration of history of no more than 6 months, erythema occupying at least one-third of the breast and pathological confirmation of invasive carcinoma.
* Hereditary cancer syndrome substudy: confirmed presence of a germline mutation known to be associated with a moderate to high lifetime risk of BC (e.g. known pathogenic variants in the genes BRCA1/2, CHEK2, TP53, PALB2) and presence of at least one malignant lesion at time of inclusion (of any origin) .
* Other substudies: no additional inclusion criteria.

Exclusion Criteria:

* Presence of a transmissible disease that can form a risk to the health of researchers or others handling the body or patient samples. This includes but is not limited to the following infectious diseases: human immunodeficiency virus (HIV), active hepatitis C virus (HCV), encephalitis of unknown cause, Creutzfeldt-Jakob disease, rabies, active malaria, active tuberculosis, active SARS-CoV-2 infection.
* Presence of any factors that could logistically or organizationally impede the study or the performance of sampling within a reasonable post-mortem time frame. This includes but is not limited to: residence of the subject at a faraway distance from the UZ Leuven hospital; residence of the subject on territory outside of Belgium; impossibility to notify the clinician confirming the death and the researchers within a reasonable time frame in case of death.

Additional exclusion criteria for the different substudies:

- ILC substudy, IBC substudy: diagnosis of a malignancy other than breast cancer in the 5 years prior to inclusion. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin and in situ cervical carcinoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2035-09 (Estimated); Study Completion 2035-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients consenting to participate in the pilot phase | Baseline
  Should be equal to or above 50%
Median time elapsed between moment of death and start of the autopsy | During autopsy
  Should be equal to or less than 12h
Median time elapsed between collection of first and last sample | During autopsy
  Should be equal to or less than 8h
Percentage of metastatic organs sampled | During autopsy
  Should be equal to or more than 75%
Percentage of samples with sufficient quality of DNA extracted | During autopsy
  A260/A280 ratio
Percentage of samples with sufficient quality of RNA extracted | During autopsy
  RNA integrity number (RIN)

SECONDARY OUTCOMES:
Concordance between TILs and clinical response to treatment | During autopsy
  Standard histopathological review
Rate of T cell exhaustion | During autopsy
  RNA sequencing
Number of mutations in each tumor lesion | During autopsy
  Whole exome sequencing
Type of mutations in each tumor lesion | During autopsy
  Whole exome sequencing
Percentage of Tumour Infiltrating Lymphocytes (TILs) | During autopsy
  Standard histopathological review

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided